CLINICAL TRIAL: NCT05757375
Title: Effects of Mulligan Ankle Taping in Volleyball Players With or Without Chronic Ankle Instability
Brief Title: Mulligan Ankle Taping on Volleyball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Özge Ecem Şenel, Research Assistant, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098
Record Dates: First submitted 2023-01-12; First posted 2023-03-07 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Chronic Ankle Instability; Mulligan
Keywords: Chronic ankle instability; Mulligan fibular taping; muscle elasticity; muscle stiffness; muscle tone

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volleyball players with Chronic Ankle Instability (Experimental): Before the taping application, the application area of all athletes will be shaved. It will be cleaned with an alcohol wipe before the application so that situations such as sweat or moisture do not reduce the effect of the banding. For taping, while the athlete lies in a supine position on a portable stretcher, the leg weight will be taken by placing the athlete's foot on the abdomen with slight knee and hip flexion. The rigid tape will be measured and cut obliquely starting approximately 2 cm anterior to the fibula and approximately 1 cm anterior to the lateral malleolus and ending in the middle of the anterior tibia region. To increase the strength of the banding, another band will be added to it. In the application, only banding will be preferred and mobilization will not be done.
  Interventions: Other: Mulligan Manuel Therapy Consept
- Volleybal players without Chronic Ankle Instability (Experimental): Before the taping application, the application area of all athletes will be shaved. It will be cleaned with an alcohol wipe before the application so that situations such as sweat or moisture do not reduce the effect of the banding. For taping, while the athlete lies in a supine position on a portable stretcher, the leg weight will be taken by placing the athlete's foot on the abdomen with slight knee and hip flexion. The rigid tape will be measured and cut obliquely starting approximately 2 cm anterior to the fibula and approximately 1 cm anterior to the lateral malleolus and ending in the middle of the anterior tibia region. To increase the strength of the banding, another band will be added to it. In the application, only banding will be preferred and mobilization will not be done.
  Interventions: Other: Mulligan Manuel Therapy Consept

INTERVENTIONS:
Other: Mulligan Manuel Therapy Consept — Mulligan ankle taping is a noninvasive, painless, low-cost, and easily applicable technique of the Mulligan manual therapy concept. It is frequently used in cases of ankle instability. In healthy people, it is a method to prevent ankle sprains.

SUMMARY:
34 volunteer professional volleyball players with (n=12) and without (n=22) CAI will include in the study. Mulligan ankle taping will apply. Measurements will take before and after the intervention. Muscle tone, stiffness, and elasticity will measure with MyotonPRO hand-held device. The static balance will measure with single leg stance test(SLST) while the eyes-closed, dynamic balance will measure with the Y balance test(YBT). Single leg hopping test(SLHT) will evaluate performance and an active position sense test will use for JPS. During the static and dynamic balance and performance tests, the ankle's confidence will be evaluated with the Visual Analog Scale (VAS). The study aimed to determine the effect of Mulligan fibular taping over the Tibialis Anterior(TA), Peroneus Longus(PL), Gastrocnemius Lateralis(GCL), and Medialis(GCM) muscles on muscle tone, stiffness, elasticity, as well as the performance, joint position sense(JPS), static and dynamic balance in female volleyball players with and without chronic ankle instability(CAI).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 15-24,
* Being a professional volleyball player,
* Training for 90 minutes at least 3 days a week,
* Turkish native speakers,
* For participants with chronic ankle instability, those with a Foot and Ankle Disability Index score below 90% and a Foot and Ankle Disability Index-Sport survey score below 75% were included.

Exclusion Criteria:

* An ankle sprain history in the last 6 weeks,
* Having a previous history of fracture in the lower extremity,
* Having bilateral chronic ankle instability,
* Pregnant athletes were excluded from the study.

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The study will be carried out on a single gender because female volleyball players experience ankle sprains more often and due to hormonal levels.
Enrollment: 34 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Myotonometric Measurement | 4 weeks
  MyotonPRO is a wireless handheld device that objectively evaluates the viscoelastic properties of muscles such as tone, stiffness, and elasticity with numerical values. It creates a mechanical effect on the subcutaneous tissue and senses the response of the tissue. The 3-millimeter probe of the device is placed 90 degrees perpendicular to the subcutaneous tissue to be measured. With the measurement, muscle tone, stiffness, and elasticity are listed numerically. Muscle tone will be calculated in hz and muscle stiffness in N/m.

SECONDARY OUTCOMES:
Single Leg Stand Test with Eyes Closed | 4 weeks
  This test, which is used to evaluate the static balance ability, is applied with bare feet on a hard and flat surface. During the test, participants are asked to close their eyes, place both hands on the opposite shoulder, and pull the untested leg to the abdomen with a 90-degree flexion angle from the hip and knee. During the test, both legs should maintain this position without touching each other. The test is started as soon as the participant's untested foot is not in contact with the ground, and is terminated when it touches the ground. The test is repeated three times for both the right and left legs and the best result is referenced.
Y Balance Test | 4 weeks
  It is a reported dynamic test with good reliability requiring strength, flexibility, and proprioception. It is a dynamic balance criterion applied to athletes and physically active people. This measurement requires a setup first. Three equal-length tapes adhere to the floor with 90°, 135°, and 135° angles between them, and a Y shape is obtained. The directions to be tested are anterior, posterolateral, and posteromedial. It is a highly reliable test to determine the risk of CABI and lower extremity injury.
Single Leg Hop Test | 4 weeks
  It is a functional performance test. This measurement requires a setup first. The 3-meter tape is placed on the floor. The athlete is asked to jump as far as possible and stay on one leg in the band. The test is invalidated when the participant touches the floor with their untested foot or takes a few more small jumps to maintain their balance after the jump. The distance from the starting level of the band to the heel contact at the end of the jump is measured. This test is repeated 3 times until a successful jump is achieved and the best result is included in the evaluation.
Joint Position Test | 4 weeks
  Joint position sense is the ability of the athlete to perceive the joint angle and repeat the same joint angle even if the extremity position changes. The active position sense test is frequently used, especially in the clinic, due to its easy application. While the test athlete's eyes are closed, he/she sits in such a way that the hip flexion angle of 90° and the knee flexion angle of 120° is achieved and the sole is in full contact with the ground. The difference between the right and left dorsiflexion angles is measured with a smartphone from the goniometer application. Dorsiflexion measurement is made by following the midline of the 5th metatarsal bone with a goniometer placed in the lateral malleolus. The athlete's ankle to be tested is passively brought to 10° dorsiflexion and returned to the starting point. Afterward, the athlete is asked to actively bring his ankle to the same angle. The test is repeated three times for both ankles. By subtracting the angle made by the athlete
Confidence in the Ankle | 4 weeks
  In order to evaluate the confidence of the athletes in the balance and performance tests, they are asked to score the confidence ratios before and after the intervention with the Visual Analogue Scale. The VAS assessment is performed for the blindfolded one-leg stance test, the Y-star balance test (anterior, posteromedial, and posterolateral aspects), and the one-leg hop tests. In order not to mislead the individual, each participant was asked, "How much was your confidence in your ankle during the test?" for each parameter. the question is asked. He is asked to show his confidence in the ankle on a 10 cm line and the distance is measured.

CONTACTS AND LOCATIONS:
Overall Officials: ÖZGE ECEM E ŞENEL, PT, Principal Investigator — İSTİNYE UNIVERSITY
Locations (1):
- Istinye University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided